CLINICAL TRIAL: NCT01412099
Title: Feasibility of a Health Promotion Program for Nontraditional College Students
Brief Title: Nutrition and Physical Activity Counseling for Nontraditional College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Lisa M. Quintiliani, PhD, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R03CA139943 (NIH); NCI-2011-00671 (Registry Identifier: NCI CLinical Trials Reporting Program)
Record Dates: First submitted 2011-08-05; First posted 2011-08-09 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Health Behavior
Keywords: Exercise; Fast Foods; Fruits; Vegetables; Beverages; Non-traditional college students; Motivational Interviewing; Peer Counselors; Cancer Prevention
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback report plus peer counseling (Experimental)
  Interventions: Behavioral: peer counseling; Behavioral: Feedback report
- Feedback report (Experimental)
  Interventions: Behavioral: Feedback report

INTERVENTIONS:
Behavioral: peer counseling — Participants receive 3 phone calls from a peer counselor to deliver counseling using motivational interviewing techniques focused on diet and physical activity behaviors over a 6 week period.
  Arms: Feedback report plus peer counseling
Behavioral: Feedback report — Participants receive a one-page printed feedback report displaying their current levels of nutrition and physical activity behaviors and tips for meeting recommended guidelines.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of two methods of delivering information about nutrition and physical activity to non-traditional college students. Participants will receive either a printed feedback report alone, or the feedback report in addition to a series of phone calls from a peer counselor. The peer counselors will provide nutrition and physical activity counseling using motivational interviewing techniques. Nutrition and physical activity outcomes will be measured for both groups and compared.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled undergraduate student at UMass Boston,
* Have completed high school,
* 24yrs old or older AND/OR part time students,
* Noncompliant in at least 1 of 4 behaviors: fruit & vegetable intake, sugar sweetened beverage intake, fast food intake, or physical activity),
* Willing to randomized into either study group,
* Be able to give informed consent.

Exclusion Criteria:

* Have any contraindications to physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
physical activity and diet behaviors (fruit and vegetable intake, sugary drink intake, and fast food intake) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Quinitiliani, PhD, RD, Principal Investigator — Boston Medical Center
Locations (1):
- University of Massachusetts Boston, Boston, Massachusetts, United States